CLINICAL TRIAL: NCT04776837
Title: Tumor Markers, Liquid Biopsies, and Patient Reported Outcomes in Metastatic Colorectal, Pancreas, Biliary, and Esophagogastric Cancers
Brief Title: Predicting Disease Progression and/or Recurrence in Cancer
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aparna Parikh, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 18-380
Record Dates: First submitted 2020-01-30; First posted 2021-03-02 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Patient Reported Outcome Measures; Colorectal Cancer; Pancreatic Cancer; Biliary Tract Cancer; Esophageal Cancer; Metastatic Cancer; Disease Progression; Survival Analysis
Keywords: Patient Reported Outcome Measures; Colorectal Cancer; Pancreatic Cancer; Biliary Tract Cancer; Esophageal Cancer; Metastatic Cancer; Disease Progression; Survival Analysis
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected serially throughout study treatment. It will be processed to separate blood cell pellet from plasma and each component will be aliquoted and frozen for subsequent analyses.
  Tissue will be obtained for next-generation sequencing from formalin fixed archival tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: * Patient-reported outcomes (e.g. symptoms, quality of life) and biomarkers compare to standard of care clinical assessments such as imaging and tumor markers in predicting the clinical outcomes (e.g. disease progression and survival)
  * Prior to starting anti-cancer therapy and at subsequent designated visits (every one month)
  * Collections include:
    * Blood sample
    * Questionnaires quality of life, mood, and symptoms
    * Tissue may be obtained for next-generation sequencing.
  Interventions: Behavioral: Observational Cohort

INTERVENTIONS:
Behavioral: Observational Cohort — Patients will be followed by collecting clinical data, biospecimens, and quality of life assessment

SUMMARY:
This is a prospective study addressing the challenge of predicting disease progression and/or recurrence in patients diagnosed with metastatic colorectal, pancreatobiliary, or esophagogastric cancer that are receiving anti-cancer therapy.

DETAILED DESCRIPTION:
This research study is evaluating how patient-reported outcomes (e.g. symptoms, quality of life) and biomarkers compare to standard of care clinical assessments such as imaging and tumor markers in predicting the clinical outcomes (e.g. disease progression and survival) in patient populations with colorectal, pancreatobiliary, or esophagogastric cancer that are receiving anti-cancer therapy Massachusetts General Hospital Cancer Center

* Patient reported outcomes will be collected through a series of self-administered questionnaires and blood draws will be used to obtain bio and tumor marker information.
* Information will also be collected from the participants electronic medical record.
* Tissue may be obtained for next-generation sequencing.
* The study will conclude after participants are no longer receiving anti-cancer therapies.
* It is expected that about 200 people will take part in this research study

ELIGIBILITY:
* Inclusion Criteria:

  * Patients must have histologically confirmed colorectal, pancreatobiliary, or esophagogastric cancer.
  * Diagnosed with metastatic disease
  * Age > 18 years.
  * Patients must be starting new line of anti-cancer therapy.
  * Patient must be English-speaking.
* Exclusion Criteria
* Unwilling or unable to participate in the study
* Non-metastatic disease
* Not starting new anti-cancer treatment
* Cognitive issues interfering with ability to participate.
* Active, unstable, untreated serious mental illness interfering with ability to participate.
* Patient does not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have histologically confirmed colorectal, pancreatobiliary, or esophagogastric cancer and receiving anti cancer treatment at Massachusetts General Hospital Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Treatment Response at 1st Scan | 6 months
  The primary outcome is treatment response (RECIST 1.1) at first scan (>1 month post-treatment start). Both response status (PR vs SD or PD [including death]) and clinical benefit status (PR or SD vs PD [including death]) will be examined. Primary analyses will compare one month change from baseline in tumor markers, MAF of the selected clonal mutation in ctDNA, and PROs (symptoms, mood, and QOL) individually and a composite score in predicting response and clinical benefit (CB) at first scan.

SECONDARY OUTCOMES:
Treatment Response at 1st Scan - Continuous Outcome | 6 months
  Change from baseline to one month for each variable (tumor markers [CEA, CA19-9], ctDNA, and PROs [symptoms, mood, QOL]) will be evaluated individually as a predictor of percent change in tumor measurements at first scan (RECIST 1.1).
Progression Free Survival - KMC | 1 year
  Estimate distributions of progression free survival using the Kaplan-Meier method.
Progression Free Survival - HR | 1 year
  Use Cox proportional hazards models to obtain hazard ratios for Progression Free Survival for change in tumor markers, ctDNA and PROs.
Overall Survival - KMC | 1 year
  Estimate distributions of overall survival using the Kaplan-Meier method.
Overall Survival - HR | 1 year
  Use Cox proportional hazards models to obtain hazard ratios for Overall Survival for change in tumor markers, ctDNA and PROs.
ROC Curves | 1 year
  The investigators will compare the predictive ability of change in tumor markers, ctDNA, and PROs in these models using time-dependent ROC curves evaluated at specific timepoints including 6 and 12 months.
PROs and Biomarkers as predictor of survival using cox proportional hazards model | 6 months
  The investigators will run multivariable Cox proportional hazards regression with purposeful selection of covariates to explore combinations of variables (change in tumor markers [CEA, CA19-9], ctDNA, and PROs [symptoms, mood, QOL]) as predictors of survival (PFS and OS).
Association between baseline PROs, biomarkers and tumor response | 6 months
  The investigators will look at correlations between baseline ctDNA levels, baseline tumor markers and baseline PRO assessments and tumor response.
Associations between baseline PROs, biomarkers, and 6-month survival outcomes | 6 months
  The investigators will look at correlations between baseline ctDNA levels, baseline tumor markers and baseline PRO assessments and 6-month survival outcomes (PFS, OS)
Sarcopenia Analysis | 1 year
  As an exploratory outcome the investigators will compare differences in demographic and clinical characteristics, PROs, and clinical outcomes, between patients with and without sarcopenia.
Skeletal Muscle Analyses | 1 year
  As an exploratory outcome the investigators will compare differences in demographic and clinical characteristics, PROs, and clinical outcomes, between patients by skeletal muscle index and density.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna R Parikh, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor- Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation